CLINICAL TRIAL: NCT00264004
Title: A Phase II, Randomised, Factorial, Double-blind Study to Investigate the Management of AZD2171-induced Hypertension and Efficacy of AZD2171 at Doses of 30 mg and 45 mg in Patients With Advanced Solid Tumours
Brief Title: Study to Investigate the Management of Hypertension and Efficacy of AZD2171 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8480C00038; EUDRACT Number 2005-003442-33
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-07

CONDITIONS: Tumors
Keywords: Advanced Solid Tumours; phase II; Hypertension; RECENTIN
MeSH Terms: conditions — Neoplasms; Hypertension | interventions — cediranib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): 30 mg AZD2171
  Interventions: Drug: AZD2171
- 2 (Experimental): 45 mg AZD2171
  Interventions: Drug: AZD2171

INTERVENTIONS:
Drug: AZD2171 — 30 mg & 45 mg oral tablet
  Other Names: Cediranib; RECENTIN™

SUMMARY:
The purpose of this study is to determine whether doses of 30 mg and 45 mg AZD2171 can be well tolerated without significant drug withdrawal when accompanied by a suitable hypertension management strategy or dose reduction.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of advanced solid tumour, which is refractory to standard therapies or for which no standard therapy exists and for which there is a rationale for the therapeutic use of a vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitor.

Exclusion Criteria:

* Prior treatment with a VEGF inhibitor
* Poorly controlled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2005-11; Primary Completion 2007-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, MD, Study Director — AstraZeneca
Locations (6):
- Germany (2):
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Nijmegen
  - Research Site, Utrecht
- Research Site, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD2171 30 mg Anti HT: AZD2171 30 mg AntiHT prophylaxis
- AZD2171 30 mg No Anti HT: AZD2171 30 mg No AntiHT prophylaxis
- AZD2171 45 mg Anti HT: AZD2171 45 mg AntiHT prophylaxis
- AZD2171 45 mg No Anti HT: AZD2171 45 mg No AntiHT prophylaxis
Period: Overall Study
Arm/Group | AZD2171 30 mg Anti HT | AZD2171 30 mg No Anti HT | AZD2171 45 mg Anti HT | AZD2171 45 mg No Anti HT
Started | 30 (Randomised) | 32 (Randomised) | 30 (Randomised) | 34 (Randomised)
Completed | 13 (Completed 12 weeks treatment) | 21 (Completed 12 weeks treatment) | 16 (Completed 12 weeks treatment) | 19 (Completed 12 weeks treatment)
Not Completed | 17 | 11 | 14 | 15
Not completed — Adverse Event | 2 | 3 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 2
Not completed — Other | 2 | 2 | 0 | 3
Not completed — Development study specific disc. crit. | 1 | 0 | 1 | 0
Not completed — Cond. under inv. worsened | 9 | 5 | 3 | 4
Not completed — Not treated | 3 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD2171 30 mg Anti HT | AZD2171 30 mg No Anti HT | AZD2171 45 mg Anti HT | AZD2171 45 mg No Anti HT | Total
Number analyzed (Participants) | 30 | 32 | 30 | 34 | 126
Age Continuous [Mean (Standard Deviation); unit: Years]
  Age | 58.1 (9.3) | 52.7 (12.9) | 56.4 (11.0) | 53.5 (11.7) | 55.175 (11.225)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 13 | 25 | 66
  Male | 18 | 16 | 17 | 9 | 60

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Requiring Temporary (>1 Day) or Permanent Withdrawal of AZD2171 Prior to Progression and Within 12 Weeks of First Dose of AZD2171
Time Frame: 12 week treatment period
Measure: Number; unit: Participants
Arm/Group | AZD2171 30 mg Anti HT | AZD2171 30 mg No Anti HT | AZD2171 45 mg Anti HT | AZD2171 45 mg No Anti HT
Number analyzed (Participants) | 30 | 32 | 30 | 34
Participants | 12 | 19 | 20 | 24

2. Primary Outcome: Proportion of Planned Dose Received During First 12 Weeks of Therapy With AZD2171
Description: Total actual dose received during the first 12 weeks prior to progression divided by the planned dose (planned dose: initial allocated dose multiplied by the number of days on study during the first 12 weeks prior to progression)
Time Frame: 12 week treatment period
Measure: Median (90% Confidence Interval); unit: Poportion of Planned Dose
Arm/Group | AZD2171 30 mg Anti HT | AZD2171 30 mg No Anti HT | AZD2171 45 mg Anti HT | AZD2171 45 mg No Anti HT
Number analyzed (Participants) | 30 | 32 | 30 | 34
Poportion of Planned Dose | 0.89 [0.62 to 1.00] | 0.88 [0.76 to 0.98] | 0.74 [0.58 to .91] | 0.79 [0.64 to 0.87]

3. Secondary Outcome: Proportion of Patients Requiring Temporary (>1 Day) or Permanent Withdrawal of AZD2171 Prior to Progression and Within 6 Weeks of First Dose of AZD2171
Time Frame: First 6 weeks of 12 week treatment period
Measure: Number; unit: Participants
Arm/Group | AZD2171 30 mg Anti HT | AZD2171 30 mg No Anti HT | AZD2171 45 mg Anti HT | AZD2171 45 mg No Anti HT
Number analyzed (Participants) | 30 | 32 | 30 | 34
Participants | 9 | 9 | 16 | 19

4. Secondary Outcome: Objective Response Rate
Description: Number of patients with complete or partial response (CR/PR), based on RECIST
Time Frame: 12 week treatment period
Measure: Number; unit: Participants
Arm/Group | AZD2171 30 mg Anti HT | AZD2171 30 mg No Anti HT | AZD2171 45 mg Anti HT | AZD2171 45 mg No Anti HT
Number analyzed (Participants) | 29 | 32 | 30 | 34
Participants | 1 | 3 | 2 | 3

5. Secondary Outcome: Best Percentage Change in Tumour Size
Description: Maximum percentage reduction or minimum percentage increase in tumour size where size is the sum of the longest diameters of the target lesions. Based on the baseline scaled ratio: ratio of the post-randomisation visit tumour size divided by the baseline tumour size.
Time Frame: Randomisation until end of treatment period
Measure: Geometric Mean (90% Confidence Interval); unit: percentage of tumor size
Arm/Group | AZD2171 30 mg Anti HT | AZD2171 30 mg No Anti HT | AZD2171 45 mg Anti HT | AZD2171 45 mg No Anti HT
Number analyzed (Participants) | 25 | 29 | 21 | 27
percentage of tumor size | -1.12 [-8.96 to 7.38] | -10.81 [-23.99 to 4.65] | -11.78 [-22.53 to 0.46] | -13.13 [-20.39 to -5.21]

ADVERSE EVENTS:
Arm/Group | AZD2171 30 mg Anti HT | AZD2171 30 mg No Anti HT | AZD2171 45 mg Anti HT | AZD2171 45 mg No Anti HT
Serious Adverse Events (participants affected / at risk) | 19/28 | 20/31 | 10/26 | 10/34
Other Adverse Events (participants affected / at risk) | 31/28 | 34/31 | 27/26 | 26/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2171 30 mg Anti HT (N=28) | AZD2171 30 mg No Anti HT (N=31) | AZD2171 45 mg Anti HT (N=26) | AZD2171 45 mg No Anti HT (N=34)
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 2 | 2
Pyrexia (General disorders) | 2 | 0 | 1 | 1
Euthanasia (General disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0
Infected Skin Ulcer (Infections and infestations) | 0 | 1 | 0 | 0
Lung Infection (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Blood Bilirubin Increased (Infections and infestations) | 0 | 1 | 0 | 0
Hepatic Enzyme Increased (Infections and infestations) | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral Pain (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 5 | 4 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Venous Thrombosis Limb (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2171 30 mg Anti HT (N=28) | AZD2171 30 mg No Anti HT (N=31) | AZD2171 45 mg Anti HT (N=26) | AZD2171 45 mg No Anti HT (N=34)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Ear Discomfort (Ear and labyrinth disorders) | 2 | 1 | 2 | 1
Hypothyroidism (Endocrine disorders) | 4 | 7 | 1 | 4
Vision Blurred (Eye disorders) | 2 | 0 | 1 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 23 | 24 | 23 | 20
Nausea (Gastrointestinal disorders) | 16 | 15 | 8 | 8
Stomatitis (Gastrointestinal disorders) | 10 | 13 | 7 | 12
Constipation (Gastrointestinal disorders) | 9 | 8 | 5 | 5
Vomiting (Gastrointestinal disorders) | 9 | 8 | 8 | 5
Abdominal Pain (Gastrointestinal disorders) | 2 | 7 | 3 | 4
Dry Mouth (Gastrointestinal disorders) | 3 | 5 | 3 | 6
Dysphagia (Gastrointestinal disorders) | 2 | 6 | 3 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 3 | 1 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 4 | 2
Ascites (Gastrointestinal disorders) | 1 | 2 | 3 | 1
Flatulence (Gastrointestinal disorders) | 0 | 3 | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Fatigue (General disorders) | 19 | 21 | 19 | 18
Pyrexia (General disorders) | 4 | 2 | 3 | 1
Asthenia (General disorders) | 1 | 3 | 1 | 1
Chills (General disorders) | 0 | 1 | 3 | 1
Mucosal Inflammation (General disorders) | 1 | 3 | 0 | 1
Oedema Peripheral (General disorders) | 3 | 3 | 2 | 1
Chest Discomfort (General disorders) | 2 | 0 | 0 | 0
Face Oedema (General disorders) | 2 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 2 | 2 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 2 | 0 | 2
Temperature Intolerance (General disorders) | 2 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 7 | 1 | 2 | 2
Cystitis (Infections and infestations) | 1 | 3 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 2 | 1 | 2
Gastrointestinal Infection (Infections and infestations) | 0 | 0 | 0 | 2
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 0 | 0
Oral Candidiasis (Infections and infestations) | 1 | 1 | 2 | 0
Rash Pustular (Infections and infestations) | 0 | 0 | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1 | 2
Viral Infection (Infections and infestations) | 0 | 2 | 0 | 0
Weight Decreased (Infections and infestations) | 8 | 5 | 3 | 3
Blood Thyroid Stimulating Hormone Increased (Infections and infestations) | 2 | 5 | 3 | 2
Alanine Aminotransferase Increased (Infections and infestations) | 2 | 3 | 2 | 0
Aspartate Aminotransferase Increased (Infections and infestations) | 1 | 1 | 2 | 0
Blood Alkaline Phosphatase Increased (Infections and infestations) | 0 | 2 | 0 | 0
Blood Bilirubin Increased (Infections and infestations) | 2 | 1 | 0 | 0
Blood Creatinine Increased (Infections and infestations) | 0 | 2 | 0 | 0
Gamma-Glutamyltransferase Increased (Infections and infestations) | 0 | 2 | 1 | 0
Transaminases Increased (Infections and infestations) | 1 | 1 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 14 | 12 | 8 | 12
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 4 | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 5 | 2
Headache (Nervous system disorders) | 7 | 6 | 2 | 9
Dizziness (Nervous system disorders) | 3 | 5 | 2 | 6
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 2 | 3 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 2 | 0
Lethargy (Nervous system disorders) | 2 | 1 | 0 | 1
Memory Impairment (Nervous system disorders) | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 0 | 1 | 2
Depression (Psychiatric disorders) | 3 | 4 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 4 | 6 | 0 | 3
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 16 | 18 | 15 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 4 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3 | 2
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 5 | 9 | 5 | 10
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 7 | 4 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 4
Nail Disorder (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 2
Hypertension (Vascular disorders) | 21 | 25 | 15 | 19
Flushing (Vascular disorders) | 0 | 2 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a Study Site, or an investigator, requests permission to publish data from this study, any such publication (including oral presentations) is to be agreed with AstraZeneca prior to publication.